CLINICAL TRIAL: NCT06652321
Title: Endothelial Side Up Inverted Femtosecond Laser Assisted DSAEK a Pilot Study
Brief Title: Endothelial Side Up Inverted Femtosecond Laser Assisted DSAEK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dar El Oyoun Hospital (Other)
Responsible Party: Principal Investigator, Tarek Haitham Ezzat Nasr, Research Associate, Dar El Oyoun Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Md-186-2021
Record Dates: First submitted 2024-08-22; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-08

CONDITIONS: Pseudophakic Bullous Keratopathy; Fuchs' Endothelial Dystrophy
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Inverted DSAEK (Experimental)
  Interventions: Procedure: Endothelial Side Up Femtosecond Laser Assisted DSAEK

INTERVENTIONS:
Procedure: Endothelial Side Up Femtosecond Laser Assisted DSAEK — The Femto LDV Z8 laser system will be set to create a 100 μm thick graft with a 7.5 mm diameter.
  The graft will be inverted, placed endothelial side up in the anterior chamber, and coated with Viscoat. A fixation ring will center the graft by holding the scleral rim with forceps.
  After cutting, the cornea should remain endothelium-up, stained with Trypan Blue, and dissected using a blunt spatula. The graft will be placed on a Busin glide and coated with Viscoat.
  A 3-4 mm corneal incision will be made, and Descemet's membrane will be marked and stripped. The graft will be inserted using the Busin glide, spreading automatically. A small air bubble will fill the anterior chamber to compress the graft for 10 minutes.

SUMMARY:
To evaluate the clinical outcomes (pos toperative best corrected visual acuity, endothelial count) and anatomical results (interface smoothness) of DSAEK with Femto LDV-prepared grafts from the endothelial side.

DETAILED DESCRIPTION:
Corneal transplantation is the most frequently performed transplant surgery worldwide, restoring visual function when corneal damage is severe. Traditionally, Penetrating Keratoplasty (PKP) was used to treat all forms of corneal blindness, but it comes with potential complications such as graft rejection, wound leaks, and astigmatism. To address these limitations, Endothelial Keratoplasty (EK) emerged as a less invasive alternative, particularly for conditions where only the corneal endothelium is compromised (e.g., Fuch's endothelial dystrophy and pseudophakic bullous keratopathy).

EK began with Posterior Lamellar Keratoplasty (PLK) and evolved through Descemet's Stripping Endothelial Keratoplasty (DSEK) and Descemet's Stripping Automated Endothelial Keratoplasty (DSAEK), which uses a microkeratome to create a thin corneal graft. DSAEK, however, results in a meniscus-shaped graft with some degree of hyperopic shift postoperatively. Another advancement, Descemet's Membrane Endothelial Keratoplasty (DMEK), uses only the donor's Descemet membrane and endothelium, providing better visual outcomes and fewer rejection risks. Despite these benefits, DMEK is technically challenging and unsuitable for some complex cases.

Ultrathin (UT) DSAEK introduced sequential microkeratome cuts, achieving graft thickness below 100 µm. This approach offers faster visual recovery and comparable refractive outcomes to DMEK, but with higher perforation risks during graft preparation. Newer graft preparation methods, such as femtosecond laser-assisted techniques, have been introduced to improve consistency, though deeper femtosecond laser cuts sometimes reduce accuracy due to laser scattering.

This study proposes using Femto LDV (Ziemer Ophthalmic Systems AG) to prepare ultrathin DSAEK grafts from the endothelial side to ensure smoother interfaces and consistent graft thickness. Previous in-vitro studies indicate that these grafts offer better endothelial protection and less damage when coated with Viscoat (sodium chondroitin sulfate 4.0%-sodium hyaluronate 3.0%) compared to basic saline solution.

Study Aim The goal of this pilot study is to evaluate the clinical outcomes (best-corrected visual acuity, endothelial cell count) and anatomical outcomes (interface smoothness) of DSAEK with Femto LDV-prepared grafts.

ELIGIBILITY:
Inclusion Criteria:

Patients with Fuchs' endothelial dystrophy Patients with bullous keratopathy secondary to intraocular surgeries, iridocorneal endothelial syndrome, or viral keratitis

Exclusion Criteria:

Bullous keratopathy secondary to glaucoma or ocular trauma Corneal stromal scarring or opacities Diseases not affecting the corneal endothelium, including corneal ectasia (e.g., keratoconus, keratoglobus, pellucid marginal degeneration) Epithelial, Bowman layer/anterior stromal, and stromal dystrophies Hypotonic eyes Retinal diseases Any type of optic atrophy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Best spectacle-corrected visual acuity | after 3 and 6 months
  Measurement Tool: Snellen chart Unit of Measure: LogMAR
Endothelial cell count using specular microscopy | after 3 and 6 months
  Measurement Tool: Specular microscopy Time Frame: After 3 months and 6 months

SECONDARY OUTCOMES:
Total central corneal thickness (CCT) | after 3 and 6 months
  Measurement Tool: Anterior Segment Optical Coherence Tomography (AS-OCT) Unit of Measure: Micrometers (µm)
Donor Corneal Endothelial Thickness (CET) | After 3 months and 6 months
  Measurement Tool: Anterior Segment Optical Coherence Tomography (AS-OCT) Unit of Measure: Micrometers (µm)

CONTACTS AND LOCATIONS:
Locations (1):
- Dar el Oyoun, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes